CLINICAL TRIAL: NCT02536937
Title: An Open-label Two-stage Pharmacokinetic and Tolerability Study of Eliglustat Tartrate Given as a Single Dose in Subjects With Mild, Moderate and Severe Renal Impairment, and in Matched Subjects With Normal Renal Function
Brief Title: A Study of the Effects of Renal Impairment on the Pharmacokinetics and Tolerability of Eliglustat Tartrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP13778; U1111-1170-3686 (Other: UTN)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GZ385660 (healthy subjects) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat
- GZ385660 (subjects with mild renal impairment) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat
- GZ385660 (subjects with moderate renal impairment) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat
- GZ385660 (subjects with severe renal impairment) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat

INTERVENTIONS:
Drug: eliglustat — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: GZ385660

SUMMARY:
Primary Objective:

To study the effect of mild, moderate, and severe renal impairment on the pharmacokinetics (PK) of eliglustat.

Secondary Objective:

To assess the tolerability of eliglustat tartrate given as a single dose in subjects with mild, moderate, and severe renal impairment in comparison with matched subjects with normal renal function.

DETAILED DESCRIPTION:
The total study duration from screening period is approximately 31 days. In stage 1, only subjects with severe renal impairment and normal renal function will be enrolled. Subjects with mild and moderate renal impairment may be enrolled in stage 2 if the results in subjects with severe renal impairment show a substantial effect of reduced renal function on pharmacokinetics.

ELIGIBILITY:
Inclusion criteria :

For renal impaired:

* Male or female subjects, between 18 and 79 years of age, inclusive.
* Body weight between 50.0 kg and 125.0 kg inclusive if male, between 40.0 kg and 110.0 kg inclusive if female, body mass index (BMI) between 18.0 and 37.0 kg/m^2, inclusive.
* Stable chronic renal impairment, as defined by Cockroft-Gault formula.
* For severe renal impairment: CrCl <30 mL/min.
* For moderate renal impairment: 30 mL/min ≤CrCl <50 mL/min.
* For mild renal impairment: 50 mL/min ≤CrCl ≤80 mL/min.

For matched subjects:

* Male or female subject, between 18 and 79 years inclusive, matched by age.
* Body weight within 15% of the body weight of the subjects with renal impairment to be matched and BMI between 18.0 and 37.0 mg/kg^2 inclusive.
* Matched by cytochrome P450 (CYP) 2D6 predicted phenotype based on genotype.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* For healthy subjects: CrCl >80 mL/min.

Exclusion criteria:

For renal impairment patients:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female) or infectious disease, or signs of acute illness.
* Active hepatitis, hepatic insufficiency.
* Acute renal failure (de novo or superimposed to pre-existing chronic renal impairment), nephrotic syndrome.
* History of or current hematuria of urologic origin that limits the subject's participation in the study.
* Subjects requiring dialysis during the study.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-hCG] blood test), breastfeeding.
* Any significant change in chronic treatment medication within 14 days before inclusion.
* P-gp inhibitors and/or inducers, CYP2D6 and/or CYP3A inducers, and strong and/or moderate CYP2D6 and/or CYP3A inhibitors. Up to one weak CYP2D6 inhibitor and/or one weak CYP3A inhibitor are allowed (as defined in The Metabolism and Transport Drug Interaction Database™ (DIDB).
* Positive result on any of the following tests: anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
* Pre-existing cardiac disease (current congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, or use of Class IA (eg, quinidine, procainamide) and Class III (eg, amiodarone, sotalol) anti-arrhythmic medications.
* Any subject with CYP2D6 indeterminate or ultra-rapid metabolizer (URM) phenotype.

For matched volunteers:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* If female, pregnancy (defined as positive β-hCG blood test), breast feeding.
* For subjects 50 years old and below: any medication (including St John's Wort) within 14 days before inclusion, or within 5 times the elimination half-life or pharmacodynamic half-life of that medication, whichever is longest, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days, and any biologics (antibody or its derivatives) within 4 months before inclusion.
* For subjects above 50 years old: any significant change in chronic treatment medication within 14 days before inclusion.
* P-gp inhibitors and/or inducers, CYP2D6 and/or CYP3A inducers, and strong and/or moderate CYP2D6 and/or CYP3A inhibitors. Up to one weak CYP2D6 inhibitor and/or one weak CYP3A inhibitor are allowed (as defined in The Metabolism and Transport Drug Interaction Database™ (DIDB).
* Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) Ab, anti-HIV1 and anti-HIV2 Ab.
* Pre-existing cardiac disease (current congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, or use of Class IA (eg, quinidine, procainamide) and Class III (eg, amiodarone, sotalol) anti-arrhythmic medications.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
- Assessment of PK parameter: Maximum plasma concentration observed (Cmax) | 3 days
- Assessment of PK parameter: Area under the plasma concentration (AUC) | 3 days

SECONDARY OUTCOMES:
Assessment of PK parameter: Area under the plasma concentration versus time curve (AUClast) | 3 days
Assessment of PK parameter: Apparent total body clearance (CL/F) | 3 days
Assessment of PK parameter: Apparent volume of distribution during the terminal phase (Vz/F) | 3 days
Assessment of PK parameter: Predicted accumulation ratio (Rac,pred) | 3 days
Assessment of PK parameter: Terminal half-life (t1/2z) | 3 days
Number of adverse events | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840004, Miami, Florida
  - Investigational Site Number 840002, Saint Paul, Minnesota
  - Investigational Site Number 840001, Knoxville, Tennessee